CLINICAL TRIAL: NCT03571386
Title: Mechanisms of Mindfulness-Based Interventions (MBIs)
Brief Title: Mechanisms of Mindfulness-based Interventions
Acronym: MBI
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Vago, Research Director; Associate Professor, Vanderbilt University Medical Center
Other Study IDs: Osher_Center_CNIM Lab
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Depression; Anxiety; Stress
Keywords: Mindfulness; Depression; Anxiety; stress
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood assays (WBA) will be used in conjunction with lipopolysaccharide (LPS)-stimulated whole blood cell cultures for detecting reliable cytokine responsivity. Introducing LPS as an in vitro stimulus to study the potential variable effect on cytokines such as TNFα gene expression in fresh whole blood as compared to fresh PBMCs or frozen PBMCs has demonstrated to be successful and with less variability than peripheral markers. The WBA uses a small sample volume (approximately 1-2 ml).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild to Moderate Depression and/or Anxiety: Patients who currently have mild to moderate severity of depression and/or anxiety symptoms are who are receiving Mindfulness-Based Cognitive Therapy (MBCT) in a group setting as standard of care will be recruited for this arm.
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy (MBCT)
- High Stress: Patients with a history of reported stress who are receiving Mindfulness-Based Stress Reduction (MBSR) in a group setting as standard of care will be recruited for this study. All patients are eligible.
  Interventions: Behavioral: Mindfulness-based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy (MBCT) — Standardized 8-week Cognitive and Behavioral Psychotherapy group with 26 hrs of in-class training and homework, along with 1 all-day retreat in which core mindfulness skills are developed
  Other Names: MBCT
  Groups: Mild to Moderate Depression and/or Anxiety
Behavioral: Mindfulness-based Stress Reduction (MBSR) — Standardized 8-week patient-centered educational approach which uses relatively intensive training in core meditation practices that teaches people how to take better care of themselves using mindfulness skills and live healthier and more adaptive lives.
  Other Names: MBSR
  Groups: High Stress

SUMMARY:
Mindfulness-based Interventions (MBIs) are a family of standardized cognitive and behavioral therapies that focus on cultivating mindfulness-related skills for improving maladaptive cognitive, emotional, and behavioral processes. MBIs have been developed for a wide range of problems, disorders, and populations and are increasingly available in a variety of health settings. This mixed methods study proposes to investigate proposed neurobiological, physiological, psycho-social-behavioral, and cognitive mechanisms by which MBIs may improve health outcomes.

DETAILED DESCRIPTION:
The state of mindfulness can be described as a form of meta-awareness in which attention is allocated to the present moment of external and internal sensory or mental experience, without reactivity, and without dwelling on any particular sensory or mental object with judgement or evaluation. Mindfulness-based Interventions (MBIs) are a family of standardized cognitive and behavioral therapies that focus on cultivating mindfulness-related skills for improving maladaptive cognitive, emotional, and behavioral processes.

MBIs have been developed for a wide range of problems, disorders, and populations and are increasingly available in a variety of health settings. Empirically supported MBIs include acceptance and commitment therapy (ACT; Hayes, Strosahl, & Wilson, 1999), dialectical behavior therapy (DBT; Linehan, 1993), mindfulness-based cognitive therapy (MBCT; Segal, Williams, & Teasdale, 2002), and mindfulness-based stress reduction (MBSR; Kabat-Zinn, 1982, 1990). Variations on these approaches, including integration of mindfulness training into individual psychotherapy from diverse perspectives, also have been described (Germer, Siegel, & Fulton, 2005). As the empirical evidence for the efficacy of these interventions continues to grow, the importance of investigating the mechanisms or processes by which they lead to beneficial outcomes is increasingly recognized. This mixed methods study proposes to investigate proposed neurobiological, physiological, psycho-social-behavioral, and cognitive mechanisms by which MBIs may improve health outcomes. Target (mechanism) engagement is expected to facilitate identification of individuals who are most likely to benefit (or not) from MBIs and further develop targeted interventions for optimization of delivery. Although there are very specific aims and hypotheses to be tested, this preliminary exploratory investigation will provide feasibility data and allow for refining existing hypotheses for larger research proposals to be submitted for extramural grant support.

ELIGIBILITY:
Across all ARMS:

* At prescreen, must be currently registered for MBCT or MBSR; at posttest, must have attended five of eight sessions for "completion".
* Must possess English language skills sufficient for providing informed consent, completing questionnaires, and understanding instructions
* Age range: 18-55
* Right-handed
* If currently taking maintenance anti-depressant and/or anti-anxiety medication, must have a "stable" regimen as indexed by no medication or dosage changes within the past three months
* No prior diagnosis of bipolar I, bipolar II, psychotic personality disorder, borderline personality disorder, and/or narcissistic personality disorder
* No current history (< 6 months) of substance abuse/dependence
* No current history (< 6 months) of regular meditation practice (>1 session/week; >10 min/session)
* No history of medical illness associated with possible changes in cerebral tissue or cerebrovasculature or with neurologic abnormality (e.g., seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, or significant head trauma, defined by loss of consciousness of ≥ 5 minutes)
* No current suicidal ideation

Eligibility for Depression & Anxiety Cohort:

Depression

* Reports having been diagnosed with non-psychotic unipolar major depressive disorder (MDD)
* ≥3 previous episodes of MDD
* Beck Depression Inventory-II (BDI-II) score between 14 and 28 (an indicator of depressive symptoms of mild to moderate severity)
* No fMRI contraindications: pregnancy, claustrophobia, or presence of a ferromagnetic object, including orthodontic braces

Anxiety:

* Reports having been diagnosed with an anxiety disorder (i.e., generalized anxiety disorder, panic disorder, specific phobia)
* Score of ≥40 on the Trait subscale of the Spielberger State-Trait Anxiety Inventory (an indicator of anxious symptoms of moderate to high severity)

Eligibility for High Stress Cohort:

- Reports of High Stress as measured by perceived Stress Scale

Eligibility for Drawing Blood:

* At least 110 pounds
* Not pregnant
* Generally healthy by self-report (i.e., free of cold and flu symptoms on the day of collection, no infections within two weeks prior to collection, no symptoms of a heart condition within six months prior to collection, no known sickle cell disease)
* Including the study draw, blood donation for clinical or research purposes within the preceding eight weeks will not exceed 550 mL
* No more than one blood draw will have occurred during the preceding week

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mindfulness-Based Cognitive Therapy or Mindfulness-based Stress Reduction program participants in an integrative health clinic
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Vago, Ph.D., Principal Investigator — Vanderbilt University Medical Center; Poppy Schoenberg, Ph.D., Principal Investigator — Vanderbilt University Medical Center; Resh Gupta, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta RS, Kujawa A, Vago DR. The neural chronometry of threat-related attentional bias: Event-related potential (ERP) evidence for early and late stages of selective attentional processing. Int J Psychophysiol. 2019 Dec;146:20-42. doi: 10.1016/j.ijpsycho.2019.08.006. Epub 2019 Oct 9. PMID 31605728
- [Background] Vago DR, Gupta RS, Lazar SW. Measuring cognitive outcomes in mindfulness-based intervention research: a reflection on confounding factors and methodological limitations. Curr Opin Psychol. 2019 Aug;28:143-150. doi: 10.1016/j.copsyc.2018.12.015. Epub 2018 Dec 27. PMID 30682701
- [Background] Vago, D. R. (2022). How meditation changes the brain: A neurophilosophical and pragmatic account. Routledge Handbook on the Philosophy of Meditation. R. Repetti. London, Routledge.
- [Background] Schuman-Olivier Z, Trombka M, Lovas DA, Brewer JA, Vago DR, Gawande R, Dunne JP, Lazar SW, Loucks EB, Fulwiler C. Mindfulness and Behavior Change. Harv Rev Psychiatry. 2020 Nov/Dec;28(6):371-394. doi: 10.1097/HRP.0000000000000277. PMID 33156156
- [Result] Gupta RS, Kujawa A, Fresco DM, Kang H, Vago DR. Mindfulness-Based Cognitive Therapy: A Preliminary Examination of the (Event-Related) Potential for Modifying Threat-Related Attentional Bias in Anxiety. Mindfulness (N Y). 2022;13(7):1719-1732. doi: 10.1007/s12671-022-01910-x. Epub 2022 Jun 1. PMID 35668874
- [Result] Gupta RS, Kujawa A, Vago DR. A Preliminary Investigation of ERP Components of Attentional Bias in Anxious Adults using Temporospatial Principal Component Analysis. J Psychophysiol. 2021 Oct;35(4):223-236. doi: 10.1027/0269-8803/a000275. Epub 2021 Feb 23. PMID 34732969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lasted through In-person and virtual 8-week MBCT courses were held in a group format with approximately 12 participants in each in-person group and 20 participants in each virtual group. Participants were recruited from the greater Nashville community through ResearchMatch, and the Osher Center for Integrative Medicine at Vanderbilt.
Period: Overall Study
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
Started | 69 | 67
Completed | 50 | 62
Not Completed | 19 | 5
Not completed — scheduling conflict | 4 | 0
Not completed — Withdrawal by Subject | 15 | 5

BASELINE CHARACTERISTICS:
Population: mild to moderate anxiety cohort was same as mild to moderate depression
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress | Total
Number analyzed (Participants) | 69 | 67 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 67 | 136
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (10) | 44 (10) | 38 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 56 | 95
  Male | 30 | 11 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race (Asian, Black/African American, White, More Than One Race) reported only
  Participants
    Asian | 3 | 1 | 4
    Black/African American | 5 | 9 | 14
    White | 58 | 52 | 110
    More Than One Race | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 69 | 67 | 136

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD (Blood-oxygen-level-dependent) Mean Signal Change From Baseline to 12 Weeks in Response to Emotional (vs. Neutral) Word Stimuli
Description: fMRI BOLD response to emotional word stimuli baseline to 12 weeks (post-MBCT). BOLD signal change (pre- to post-MBCT) is estimated from the contrast of emotional word vs neutral words, and extracted from voxels within the fronto-parietal and default mode areas at baseline and 12-weeks. Significant Voxel-wise BOLD activity is reported using z-scores from peak voxels. A mean score was calculated based on z-score and SD of 2 in the context of reporting fMRI BOLD data here. Z-scores is a statistical measure that describes how many standard deviations a data point (e.g., a voxel's signal) is from the mean of the distribution of that signal. The higher the reported mean, the less likely the observed activation is due to chance, thus indicating more significant activity or activation in that particular brain region.
Time Frame: Baseline to 12 weeks
Population: Only 16 participants in Mild to moderate depression and/or anxiety participated in fMRI data collection. Participants in the "High Stress" Arm/Group were not assessed using fMRI and the subgroup was smaller given financial constraints.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
Number analyzed (Participants) | 16 | 0
units on a scale
  BOLD - Right Frontopolar Cortex | | 2.315 (.5) |
  BOLD - Right Dorsolateral PFC | | 2.13 (.5) |
  BOLD - Left Precuneus | | -2.255 (.5) |

2. Secondary Outcome: Amplitude of P1 Event-related Potentials (ERP) in Response to Threat (vs. Neutral) Face Cues Pre- to Post-MBCT
Description: P1 Evoked event-related electrical potentials (ERP) amplitudes elicited from specific emotional threat vs. neutral stimuli were primary outcome. An 80-150 ms search window at EEG electrode P8 was used to identify the P1 peak, & mean value around peaks (50 ms) was exported for analysis. Mean P1-Cue amplitudes were analyzed pre- to post-MBCT to determine the effects of time (pre to post-MBCT), emotion (angry vs. happy), and congruency (congruent vs. incongruent). Mean P1-Cue amplitudes in microvolts and SD for each condition are summarized below.
Time Frame: Baseline to 12 weeks (pre- to post-MBCT)
Population: only depression/anxiety cohorts participated in ERP analyses. High stress group was not analyzed using ERP analyses
Measure: Mean (Standard Deviation); unit: mean amplitude in microvolts & SD
Groups:
- Mild to Moderate Depression and/or Anxiety: Patients who currently have mild to moderate severity of anxiety symptoms are who are receiving Mindfulness-Based Cognitive Therapy (MBCT) in a group setting as standard of care will be recruited for this arm.
  Mindfulness-based Cognitive Therapy (MBCT): Standardized 8-week Cognitive and Behavioral Psychotherapy group with 26 hrs of in-class training and homework, along with 1 all-day retreat in which core mindfulness skills are developed
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
Number analyzed (Participants) | 50 | 0
mean amplitude in microvolts & SD
  Mean amplitude (uv) and standard deviations for Angry Cues pre-MBCT | 2.62 (2.83) |
  Mean amplitude (uv) and standard deviations for Angry Cues post-MBCT | 2.60 (2.74) |
  Mean amplitude (uv) and standard deviations for Happy Cues pre-MBCT | 2.68 (2.81) |
  Mean amplitude (uv) and standard deviations for Happy Cues post-MBCT | 2.58 (2.73) |
  Mean amplitude (uv) and standard deviations for Angry Congruent Cues pre-MBCT | 1.19 (2.32) |
  Mean amplitude (uv) and standard deviations for Angry Congruent Cues post-MBCT | .87 (1.97) |
  Mean amplitude (uv) and standard deviations for Angry Incongruent Cues pre-MBCT | 1.16 (2.30) |
  Mean amplitude (uv) and standard deviations for Angry Incongruent Cues post-MBCT | .61 (2.24) |
  Mean amplitude (uv) and standard deviations for Happy Congruent Cues pre-MBCT | 1.19 (2.42) |
  Mean amplitude (uv) and standard deviations for Happy Congruent Cues post-MBCT | .64 (2.22) |
  Mean amplitude (uv) and standard deviations for Happy Incongruent Cues pre-MBCT | 1.14 (2.15) |
  Mean amplitude (uv) and standard deviations for Happy Incongruent Cues post-MBCT | .65 (2.11) |

3. Secondary Outcome: Response Time to Probes as a Function of Emotion and Congruency in the Dot Probe Task
Description: Effects of time (pre-MBCT versus post-MBCT), emotion (angry versus happy), and congruency (congruent probes versus incongruent probes) on reaction time (RT) was measured in mild to moderate depression/anxiety group.
Time Frame: Baseline to ~12 weeks
Population: Only Mild to moderate depression and/or anxiety cohort who completed MBCT was analyzed for the dot-probe task. Data for this assessment was not collected from participants in the "High Stress" Arm
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
Number analyzed (Participants) | 50 | 0
milliseconds
  RT to probes congruent with angry emotional stimuli pre-MBCT | unit of measure: mean RT & SE) | 303.50 (1.2) |
  RT to probes congruent with angry emotional stimuli post-MBCT | unit of measure: mean RT & SE | 298.30 (1.2) |
  RT to probes incongruent with angry emotional stimuli pre-MBCT | unit of measure: mean RT & SE | 304.51 (1.3) |
  RT to probes incongruent with angry emotional stimuli post-MBCT | unit of measure: mean RT & SE | 301.29 (1.5) |
  RT to probes congruent with happy emotional stimuli pre-MBCT | unit of measure: mean RT & SE | 301.47 (1.4) |
  RT to probes congruent with happy emotional stimuli post-MBCT | unit of measure: mean RT & SE | 297.5 (1.3) |
  RT to probes incongruent with happy emotional stimuli pre-MBCT | unit of measure: mean RT & SE | 304.22 (1.2) |
  RT to probes incongruent with happy emotional stimuli post-MBCT | unit of measure: mean RT & SE | 301.38 (1.1) |

4. Other Pre Specified Outcome: Self-report Psychological Measures of Anxiety and Stress Pre- to Post-Mindfulness Training
Description: The Depression & Anxiety Stress Scale (DASS-Anxiety) (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess symptoms of fear and autonomic arousal. Items are rated on a 4-point scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. The DASS-Depression is a 7-item measure designed to assess dysphoric mood. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance.
Time Frame: Baseline to ~12 weeks pre- to post-MBCT (depression/anxiety cohort)
Population: Only 50 of the Depression and anxiety cohort who completed MBCT were tested on DASS-Anxiety and DASS-Depression pre/post MBCT; High Stress cohort was tested using the Perceived Stress Scale and reported in other outcomes
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
Number analyzed (Participants) | 50 | 0
Score on a scale
  DASS-D scores pre- to post-MBCT | Mean change scores, (SE) | 7.96 (1.41) |
  DASS-A mean change pre- to post-MBCT | mean change, (SE) | 3.68 (1.28) |

5. Other Pre Specified Outcome: Self-report Psychological Measures of Stress Pre- to Post-Mindfulness Training
Description: The Perceived Stress Scale (PSS-14) is a 14-item scale, with a total range from 0 (no symptoms) to 56 (highest severity) Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance.
Time Frame: Baseline to ~12 weeks pre- to post-MBSR (high stress cohort)
Population: Only the High Stress cohort was tested using the Perceived Stress Scale (PSS-14); Depression and anxiety cohort was tested on DASS-Anxiety and DASS-Depression and reported in other outcomes
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
Number analyzed (Participants) | 0 | 62
Score on a scale |  | -7.4 (2.3)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Description: Definitions for adverse events do not differ from clinicaltrials.gov
Arm/Group | Mild to Moderate Depression and/or Anxiety | High Stress
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/67
Other Adverse Events (participants affected / at risk) | 0/69 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03571386/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03571386/ICF_001.pdf